CLINICAL TRIAL: NCT02758769
Title: Long-Term Outcomes With Abatacept In Biologic Treatment-Naive Rheumatoid Arthritis Patients In Japanese Clinical Practice Settings
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-574
Record Dates: First submitted 2016-04-14; First posted 2016-05-02 (Estimated); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole Blood

GROUPS / COHORTS (1):
- ORENCIA with Exposure: ORENCIA with Exposure
  Interventions: Biological: ORENCIA Subcutaneous Injection

INTERVENTIONS:
Biological: ORENCIA Subcutaneous Injection
  Other Names: Abatacept

SUMMARY:
The purpose of this study is to examine the effectiveness and safety of the abatacept administration in biologic-naïve rheumatoid arthritis patients who have moderate disease activity despite treatments with conventional synthetic disease modified anti-rheumatic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with RA who meet the 2010 American College of Rheumatology / European League against Rheumatisms (ACR/EULAR) RA Classification Criteria
* Patients with RA with a moderate disease activity (SDAI: > 11 and 26)
* Biologic-naive patients with treatment history csDMARDs
* Patients who meet the following criteria by hematological examination:

  * Peripheral white blood cell count: 4,000/mm3
  * Peripheral lymphocyte count: 1,000/mm3
  * Blood β-D-glucan negative
* Patients who understand the investigator's explanation of study procedures and have given voluntary written consent to participate in this study
* Patients initiated with abatacept at per their physician's therapeutic decision

Exclusion Criteria:

* Past history of hypersensitivity to the components of the abatacept preparation
* Disease complications from a comorbidity
* Active infectious disease
* Been judged by the investigator or the co-investigator as being inappropriate

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Percentage of achievement in simplified disease activity index (SDAI) remission after administration of abatacept | 52 Weeks

SECONDARY OUTCOMES:
Percentage of achievement in low disease activity by simplified disease activity index (SDAI). | 52 Weeks
Change in the percentage of disease activity category by simplified disease activity index(SDAI) | 0 Months, 1 Month, 6 Months, 12 Months, 18 Months, 24 Months, 30 Months, 36 Months, 42 Months, 48 Months, 54 Months and 60 Months
Change in the percentage of disease activity category by clinical disease activity index(CDAI) | 0 Months, 1 Month, 6 Months, 12 Months, 18 Months, 24 Months, 30 Months, 36 Months, 42 Months, 48 Months, 54 Months and 60 Months
Change in the percentage of disease activity category by disease activity score with 28 joint counts - erythrocyte sedimentation rate (DAS28-ESR) | 0 Months, 1 Month, 6 Months, 12 Months, 18 Months, 24 Months, 30 Months, 36 Months, 42 Months, 48 Months, 54 Months and 60 Months
Change in the percentage of disease activity category by disease activity score with 28 joint counts creactive protein (DAS28-CRP) | 0 Months, 1 Month, 6 Months, 12 Months, 18 Months, 24 Months, 30 Months, 36 Months, 42 Months, 48 Months, 54 Months and 60 Months
Change in simplified disease activity index(SDAI) | 0 Months, 1 Month, 6 Months, 12 Months, 18 Months, 24 Months, 30 Months, 36 Months, 42 Months, 48 Months, 54 Months and 60 Months
Change in clinical disease activity index(CDAI) | 0 Months, 1 Month, 6 Months, 12 Months, 18 Months, 24 Months, 30 Months, 36 Months, 42 Months, 48 Months, 54 Months and 60 Months
Change in disease activity score with 28 joint counts - erythrocyte sedimentation rate (DAS28-ESR) | 0 Months, 1 Month, 6 Months, 12 Months, 18 Months, 24 Months, 30 Months, 36 Months, 42 Months, 48 Months, 54 Months and 60 Months
Change in disease activity score with 28 joint counts Creactive protein (DAS28-CRP) | 0 Months, 1 Month, 6 Months, 12 Months, 18 Months, 24 Months, 30 Months, 36 Months, 42 Months, 48 Months, 54 Months and 60 Months
Change in Anti-citrullinated protein antibodies (ACPA) | 0 Months, 1 Month, 6 Months, 12 Months, 18 Months, 24 Months, 30 Months, 36 Months, 42 Months, 48 Months, 54 Months and 60 Months
Change in Rheumatoid factors (RF) | 0 Months, 1 Month, 6 Months, 12 Months, 18 Months, 24 Months, 30 Months, 36 Months, 42 Months, 48 Months, 54 Months and 60 Months
Survival rate | 0 Months, 1 Month, 6 Months, 12 Months, 18 Months, 24 Months, 30 Months, 36 Months, 42 Months, 48 Months, 54 Months and 60 Months
Hospitalization rate | 0 Months, 1 Month, 6 Months, 12 Months, 18 Months, 24 Months, 30 Months, 36 Months, 42 Months, 48 Months, 54 Months and 60 Months
Number of occurrences of rheumatoid arthritis related surgery | 0 Months, 1 Month, 6 Months, 12 Months, 18 Months, 24 Months, 30 Months, 36 Months, 42 Months, 48 Months, 54 Months and 60 Months
Persistence rate of Abatacept treatment | 0 Months, 1 Month, 6 Months, 12 Months, 18 Months, 24 Months, 30 Months, 36 Months, 42 Months, 48 Months, 54 Months and 60 Months
Reasons for discontinuation of Abatacept treatment | 0 Months, 1 Month, 6 Months, 12 Months, 18 Months, 24 Months, 30 Months, 36 Months, 42 Months, 48 Months, 54 Months and 60 Months
Change in Japanese Health Assessment Questionnaire | 0 Months, 1 Month, 6 Months, 12 Months, 18 Months, 24 Months, 30 Months, 36 Months, 42 Months, 48 Months, 54 Months and 60 Months
Change in European Quality of Life 5 Dimension Questionnaire | 0 Months, 1 Month, 6 Months, 12 Months, 18 Months, 24 Months, 30 Months, 36 Months, 42 Months, 48 Months, 54 Months and 60 Months
Change in Pain visual analog scale | 0 Months, 1 Month, 6 Months, 12 Months, 18 Months, 24 Months, 30 Months, 36 Months, 42 Months, 48 Months, 54 Months and 60 Months
Change in General visual analog scale | 0 Months, 1 Month, 6 Months, 12 Months, 18 Months, 24 Months, 30 Months, 36 Months, 42 Months, 48 Months, 54 Months and 60 Months
Change in PRO parameters defined in IORRA registry (JMAJ 2009 52 (1) 54-56) | 0 Months, 1 Month, 6 Months, 12 Months, 18 Months, 24 Months, 30 Months, 36 Months, 42 Months, 48 Months, 54 Months and 60 Months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Japan (2):
  - Local Institution - 0001, Minato-ku, Tokyo
  - Local Institution, Minato-ku, Tokyo

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm